CLINICAL TRIAL: NCT01877317
Title: Study of SelfFit App for Hearing Loss Diagnostics Based on Threshold Measurements Through In-situ Audiometry and Adjustment of Hearing Device Amplification Parameters in Agreement With Prescriptive Formulas as NAL-NL1,DSL-i/o
Brief Title: Study of SelfFit Mobile Medical App for Hearing Loss Diagnostics and Hearing Device Fitting / Fine Tuning
Acronym: SelfFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Two Pi Signalprocessing Applications GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZIT-653820; NL44209.018.13 (Other: Dutch Medical Ethics Review Committee)
Record Dates: First submitted 2013-05-28; First posted 2013-06-13 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Mild to Moderate Sensorineural Hearing Loss
Keywords: Audiology; hearing loss; hearing healthcare; mobile app; hearing aid fitting; audiometry; audiogram
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SelfFit adjusted hearing device (Experimental): Hearing impaired people with mild to moderate sensorineural hearing loss (PTA124<50 dB) in the test ear compare the performance of their hearing aids adjusted through SelfFit mobile medical App (I-Pad) with the performance of their hearing aids adjusted through conventional audiogram-based fitting.
  Interventions: Device: SelfFit adjusted hearing device

INTERVENTIONS:
Device: SelfFit adjusted hearing device — Comparison of threshold measurements through in-situ audiometry with full diagnostic audiometry; Comparison of First-Fit based on SelfFit-formula with conventional fitting formula NAL-NL1 (IG-measurements; Speech intelligibility with First fit of SelfFit; Speech intelligibility with Final fit of SelfFit; Comparison of fine tuning through SelfFit (Final fit) with First fit; Comparison of Final fit with Traditional fit (conventional fitted hearing aid of the test person)
  Other Names: User-fitted hearing device; hearing device fitting software; home-fitting tool for hearing devices

SUMMARY:
The purpose of this clinical study is to validate the comparability of prescription formula fitting of hearing aids based on full diagnostic audiometry and SelfFit interactive fitting of hearing aids based on hearing loss screening (mild to moderate hearing losses) using in-situ audiometry, provided and executed through the mobile medical app.

DETAILED DESCRIPTION:
The technology utilized within the mobile medical App is partially described in the US patent application US2011/0002490A1. The app is to be used in combination with a hearing aid to deliver the output and targets accurate individual acoustical amplification for effective compensation of a users hearing loss.

The electronic circuitry incorporating the digital signal processing algorithms - dynamic range compression, noise reduction - is providing the acoustical amplification according to parameters (acoustical gain, compression ratio, time constants) calculated through the App on base of in-situ hearing loss diagnostics (pure tone audiometry, loudness scaling). Within the study, amplification parameters will be transmitted to the prototyped device through a prototyped audio streaming box.

Individual audiogram represents hearing thresholds (softest audible sounds) at different frequencies. At least two test frequencies are used involving one in the lower region of device's bandwidth (such as 750 Hz) and one in the higher region of the device's bandwidth (such as 2 kHz). Hearing thresholds are assessed by presenting pure tones of different known levels (SPL) to the user and the thresholds for each of the test frequencies are determined according to the user response to a verbally formulated question (how many tones did you hear?) and multiple choice answer buttons (0, 1, or 2).

Second hearing loss characteristic obtained by the app. is the personal loudness scaling. By presenting a band-limited noise stimuli and collecting the user response about perceived loudness level Medical Mobile App calculates dynamic range of users hearing at given frequency.

The calculation of optimal amplification parameters is performed by App using a proprietary "fitting formula" derived from scientific data.

Final adjustment of amplification parameters called fine tuning is performed while presenting the user with realistic acoustical environment during operation of the hearing device. Fine tuning relates to slight changes of the parameters initially obtained by the "fitting formula". The acoustical signals are presented using audio streaming through the hearing aid. In particular the presented signals include "speech in quiet" and "speech in background noise". Presented speech signal is composed from two or more sources that are processed with different signal processing parameters. During the presentation of the speech signal App presents the speech source visually as two or more speakers. The user is asked to provide his listening preference by choosing the preferred speaker. The signal processing parameters relating to the preferred sound are used for final adjustment of hearing device.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss at the better ear between 35dB and 50dB (PTA1/2/4)
* Active lifestyle
* No language problems
* No medical contra-indications
* Age: between 18 and 75 years
* About 50% experienced users and 50% new users
* Willing to participate in the trial with one three hour visit to the AMC.

Exclusion Criteria:

* Conductive hearing loss in the middle ear
* Severe hearing loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hearing threshold | June - July 2013 (up to 2 months)
  Applicability of in-situ audiometry:
  Comparison of pure tone audiometry outcomes: conventional full diagnositic and SelfFit in-situ audiometry

SECONDARY OUTCOMES:
Speech intelligibility - First Fit | June - July 2013 (up to 2 months)
  Quality of First-Fit:
  Comparison speech audiometry with CVC words @ 55/65/75 db SPL in conventionally adjusted hearing aid and SelfFit adjusted hearing aid

OTHER OUTCOMES:
Speech intelligibility - Final Fit | June - July 2013 (up to 2 months)
  Quality of Final-Fit:
  Comparison speech audiometry with CVC words @ 55/65/75 db SPL in conventionally adjusted hearing aid and SelfFit adjusted hearing aid

CONTACTS AND LOCATIONS:
Overall Officials: Wouter A Dreschler, Prof.dr.ir., Principal Investigator — Department of Clinical & Experimental Audiology of the Academic Medical Centre in Amsterdam
Locations (1):
- Department of Clinical & Experimental Audiology of the Academic Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No